CLINICAL TRIAL: NCT02554227
Title: Verification and Progress of Cytokine Profiles and suPAR for the Discrimination of Infectious and Non-infectious, Degenerative Diseases of the Spine
Brief Title: Cytokine Profiles and suPAR in Spondylodiscitis
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Ayla Yagdiran, Dr.med., University of Cologne
Other Study IDs: Uni-Köln_11_2014
Record Dates: First submitted 2015-09-15; First posted 2015-09-18 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Spondylodiscitis
Keywords: Spondylodiscitis; erosive osteochondrosis; infection; cytokine profiles; lumbar, thoracic spine; suPAR
MeSH Terms: conditions — Discitis; Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bio-Plex Pro Human Cytokine Group I 27-plex Assay (IL-1β, IL-1ra, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-10, IL-12 (p70), IL-13, IL-15, IL-17, FGF basic, Eotaxin, G-CSF, GM-CSF, IFN-γ, IP-10, MCP-1, MIP-1α, MIP-1β, PDGF-BB, RANTES, TNF-α, VEGF), suPAR (soluble urokinase-type plasminogen activator receptor)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Spondylodiscitis: vertebral osteomyelitis, erosive osteochondrose
  Interventions: Other: Cytokine Profile and suPAR

INTERVENTIONS:
Other: Cytokine Profile and suPAR — Routine blood collection will be carried out directly before surgery and also during the stationary hospitalization on day 4 and day 10. Additional blood collection will be done after 6 weeks and 3 months during the follow-up.

SUMMARY:
Spondylodiscitis is an infectious disease of the intervertebral discs and adjacent vertebral bodies, which often has a protracted progression. Diagnosis is frequently delayed because of the unspecific pathology and a lack of specific infection markers. However, an early diagnosis is fundamental to prevent long periods with symptoms including extensive back pain and progressive and destructive changes of the spine.

Cytokines can be helpful to extend the knowledge about diverse biological processes. Furthermore, they are a promising category of biomarkers that are already present in the early phases of developing diseases. Currently, little is known about the participation of cytokines in Spondylodiscitis. The aim of this study is to establish a non-invasive method to improve the diagnosis of spondylodiscitis. Therefore, blood and tissue samples will be analyzed at different time points for the concentration of specific cytokines to select potential marker cytokines via a Multiplex Assay and suPAR (soluble urokinase-type plasminogen activator receptor) via ELISA. After successful identification of the biomarkers cytokines and suPAR, verification of the results will be done by expression analysis of cytokine-producing cells.

The potential of such a diagnostic method lies in reducing medical costs and preventing extensive pain and structural changes of the spine.

Experimental research will be performed with the approval of the ethic committee of the medical faculty of the University of Cologne.

DETAILED DESCRIPTION:
Spondylodiscitis is a primary infection of the intervertebral discs with secondary infection of the adjacent end-plates and vertebral bodies. It is relatively rare with an incidence of 2.4:100.000 and three times more common among men. The process of infection, which is commonly creeping, leads to a destruction of the vertebral bodies and production of abscesses, which can cause neurological deficits.

Clinical symptoms, especially in the early stages, are uncommon. Patients suffer from unspecific back pain and fever occurs only in 50% of all cases. Currently, markers used including leucocyte count, erythrocyte sedimentation rate (ESR) and C-reactive protein (CRP) are also unspecific.For this reason of that several weeks may elapse between the first signs of symptoms and the final diagnosis of spondylodiscitis. Therefore, the identification of the pathogen is indispensable for an effective antibiotic therapy.

Spinal infections are generally monomicrobial, frequently with a haematogenous source. Therefore, blood cultures can be used for identifying the pathogens. In case of negative blood cultures, the pathogens can be identified by invasive methods such as percutaneous punch biopsy or CT-guided fine needle aspiration. Despite biopsies, the pathogen can only be identified in two out of three patients. Failures of pathogen identification are mainly due to previous systemic antibiotic treatment. As a consequence, diagnosis is often based on medical imaging methods (CT, MRT, PET, radiograph, skeletal scintigraphy). The disadvantage of these methods is that structural changes of the spine must occur to become visible.

Treatment of an advanced spondylodiscitis consists of removal of the necrotic tissue, stabilization of the affected vertebral bodies and concomitant antibiotic therapy. Randomized studies for the duration of antibiotic treatments have not been published as yet. Current recommendations are between 6 to 12 weeks. For evaluating the therapy response only the clinical improvement and the CRP value are used. The mean period of stay in the hospital is about 49 days.

The goal is to establish a non-invasive method which allows discrimination of infectious and non-infectious diseases to improve the diagnosis of spondylodiscitis. For that purpose, blood and tissue samples from patients with spondylodiscitis and erosive osteochondrosis will be collected and analyzed for their cytokine and suPAR concentration. Erosive osteochondrosis is a non-infectious, degenerative disease of the spine with similar surgical treatment. Thus, it is an optimal reference group. Nevertheless, erosive osteochondrosis includes special types, called modic type I-III. Because modic type I is associated with an immune response caused by repeated traumata of the spine this modic type will be excluded from the study.

Cytokines are messengers, which are present in blood and all tissues, regulating the immune response. In this study, the goal is to assess if cytokine profiles and suPAR contribute to the discrimination of infectious and non-infectious spondylodiscitis and if this could be verified by the characterization of the cytokine-producing cells. Furthermore, the investigators want to analyze the therapy response by measuring the cytokine and suPAR profiles.

Routine blood collection will be carried out directly before surgery and also during the stationary hospitalization on day 4 and day 10. Additional blood collection will be done after 6 weeks and 3 months during the follow-up. At each time point serum and plasma will be used for the study to determine the cytokine and suPAR concentration and expression of the cytokine-producing cells. Necrotic tissue, which is removed during the surgery, will be analyzed microbiologically as well as pathologically. Parts of this tissue will also be used for the determination of cytokines. Further blood samples will be collected when a patient appears again in the Department of Orthopaedic Surgery and Traumatology because of treatment and therapy of a re-infection. A minimum of 15 patients per group - control group (erosive osteochondrosis modic type II-III) and spondylodiscitis - will be included in this study. Both groups should be homogeneous in sex and age distribution.

There will be no additional pain or complications for the patients participating in this study. All samples will be collected for a period of about one year and stored at -80°C. Afterwards, the blood and tissue samples will be analyzed for potential marker suPAR via ELISA and cytokines by using a Multiplex Assay. Furthermore, results will be linked to anamnesis to detect potential correlations. Specific correlations can indicate a diagnostic and perhaps a prognostic value of the measured cytokines and suPAR.

ELIGIBILITY:
Inclusion Criteria:

* Existence of an informed consent
* Legal competence of the patient
* Lumbar and thoracic spine pathology with an indication of spondylodiscitis or rather erosive osteochondrosis
* Surgical stabilization of the affected lumbar and thoracic vertebral bodies and a removal of the affected intervertebral discs

Exclusion Criteria:

• Patients with autoimmune diseases, chronic infections (HIV, hepatitis B and C), acute infections of other parts besides the spine and active cancer diseases

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with spondylodiscitis, erosive osteochondrosis
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with high cytokine and suPAR profiles as a measurement for the diagnosis of spondylodiscitis | Change from Baseline in different Cytokine and suPAR profiles to 3 month after surgery
  different cytokine and suPAR profiles between groups

SECONDARY OUTCOMES:
Number of patients with high cytokine and suPAR profiles as a measurement for the diagnosis of vertebral osteomyelitis | Change from Baseline in different Cytokine and suPAR profiles to 3 month after surgery
  cytokines and suPAR in tissues/cells

CONTACTS AND LOCATIONS:
Overall Officials: Jan Siewe, Dr. med., Principal Investigator — University Hospital, Department of Orthopaedic Surgery and Traumatology,
Locations (1):
- Studienzentrum Orthopädie & Unfallchirurgie, Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Scharrenberg JS, Yagdiran A, Brinkmann J, Brune M, Siewe J, Jung N, Mahabir E. The diagnostic value of soluble urokinase-type plasminogen activator receptor (suPAR) for the discrimination of vertebral osteomyelitis and degenerative diseases of the spine. J Orthop Surg Res. 2019 Nov 14;14(1):367. doi: 10.1186/s13018-019-1420-6. PMID 31727136